CLINICAL TRIAL: NCT05355415
Title: Adaptive Optics Imaging of Outer Retinal Diseases
Status: Recruiting | Type: Observational
Sponsor: Food and Drug Administration (FDA) (U.S. Federal Agency)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Daniel X. Hammer, Deputy Director, Division of Biomedical Physics, Food and Drug Administration (FDA)
Other Study IDs: 2019-CDRH-074
Record Dates: First submitted 2022-04-19; First posted 2022-05-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Retinal Degeneration; Age-Related Macular Degeneration; Retinitis Pigmentosa; Hydroxychloroquine Retinopathy; Usher Syndromes; Late-Onset Retinal Degeneration; Cone Dystrophy; Cone Rod Dystrophy; Rod Cone Dystrophy; Rod Dystrophy
MeSH Terms: conditions — Retinal Degeneration; Macular Degeneration; Retinitis Pigmentosa; Usher Syndromes; Late-Onset Retinal Degeneration; Cone Dystrophy; Cone-Rod Dystrophies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Outer retinal disease: Subjects with outer retinal disease affecting the photoreceptor-retinal pigment epithelium complex will be classified by clinical exam by an experienced retina specialist. Outer retinal disease subjects will undergo adaptive optics (AO) imaging of several macular locations.
  Interventions: Device: Adaptive optics imaging
- Healthy control: Age-matched healthy control subjects will undergo the same AO imaging procedures as subjects with outer retinal diseases.
  Interventions: Device: Adaptive optics imaging

INTERVENTIONS:
Device: Adaptive optics imaging — Adaptive optics scanning laser ophthalmoscopy (AOSLO) and adaptive optics - optical coherence tomography (AO-OCT) retinal imaging

SUMMARY:
The objective of the study is to collect adaptive optics (AO) retinal images from human subjects with outer retinal diseases (diseases of the outer retina including photoreceptor, retinal pigment epithelium (RPE), basement membrane or choroidal pathologies) to develop new diagnostic methods, biomarkers, and clinical endpoints.

DETAILED DESCRIPTION:
Objective: The objective of the study is to collect adaptive optics (AO) retinal images from human subjects with outer retinal diseases (diseases of the outer retina including photoreceptor, retinal pigment epithelium (RPE), basement membrane or choroidal pathologies) to develop new diagnostic methods, biomarkers, and clinical endpoints.

Study Population: Up to fifty (50) healthy volunteers without eye disease (Cohort 1) and up to fifty (50) affected participants with any type of outer retinal disease (Cohort 2) will be enrolled.

Design: This is a longitudinal study protocol where participants will be imaged with investigational multimodal AO (mAO) retinal imaging systems that include optical coherence tomography (OCT) and scanning laser ophthalmoscopy (SLO) channels over three years. High resolution OCT and SLO videos will be collected while the instruments automatically detect and correct for image distortion caused by ocular aberrations. In general, videos of different retinal cellular structures will be acquired from several retinal locations using various imaging modes.

Outcome Measures: The primary outcomes for this protocol are development of new diagnostic methods and disease biomarkers, investigation of cellular morphological and functional changes due to various outer retinal diseases, and development of new AO clinical endpoints for novel therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Are 21 years of age or older,
2. Have the ability to cooperate with instructions during adaptive optics imaging (similar to instructions given during a clinical eye exam),
3. Have the ability to understand and sign an informed consent. (Non-English speaking participants will not be enrolled into the study), and
4. Have been diagnosed with outer retinal disease or condition (Cohort 2).

Exclusion Criteria:

1. Have a condition which prevents adequate images from being obtained (e.g. unstable fixation or media opacity),
2. Have visual correction outside of the range +4 diopters (D) to -8 D,
3. Have a history of adverse reaction to mydriatic drops,
4. Have a predisposition to (i.e., narrow iridocorneal angle) or any history of acute angle closure glaucoma (AACG), or
5. Are working under the direct supervision of Drs. Hammer, Cukras and Liu, or any of the NIH/NEI AIs.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All study participants will be recruited from the NIH patient population.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-27 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
Photoreceptor (PR) density | PR density will be calculated once at the AO imaging session in which PRs are the target.
  PR density will be calculated at specific retinal eccentricities from cells counted in average AO-OCT volumes or average AOSLO frames.
Retinal pigment epithelial (RPE) cell density | RPE cell density will be calculated once at the AO imaging session in which RPE cells are the target.
  RPE cell density will be calculated at specific retinal eccentricities from cells counted in average AO-OCT volumes.
RPE cell organelle motility | RPE motility will be calculated once at the AO imaging session in which RPE cells are the target. For the reproducibility portion of the study, RPE organelle motility will be quantified three times separated by 1-2 weeks.
  RPE cell organelle motility will be calculated from the decorrelation time constant for cells segmented from a sequence of AO-OCT volumes.
PR cell function | PR function will be calculated once at the AO imaging session in which PR cells are stimulated. For the reproducibility portion of the study, PR cell function will be quantified three times separated by 1-2 weeks.
  Photoreceptor cell (cone) function will be measured from phase changes between inner segment - outer segment junction and cone outer segment tip signals in a sequence of AO-OCT volumes collected during visible light stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel X Hammer, Ph.D., Principal Investigator — Food and Drug Administration (FDA)
Locations (2):
- United States (2):
  - NIH Clinical Center, Bethesda, Maryland
  - Food and Drug Administration, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: Yes
De-identified AO images will be shared with external academic collaborators.
Time Frame: For the duration of the study.
Access Criteria: Available upon request.

DOCUMENTS (2):
  • Study Protocol (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT05355415/Prot_004.pdf
  • Informed Consent Form (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT05355415/ICF_003.pdf